CLINICAL TRIAL: NCT03104816
Title: The Effectiveness of IV/PO Acetaminophen in the Perioperative Period in Reducing Opiate Use After Lumbar Spine Fusion: a Prospective, Randomized Controlled Trial
Brief Title: The Effectiveness of IV/PO Acetaminophen in the Perioperative Period in Reducing Opiate Use After Lumbar Spine Fusion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Could not get an approval from Department Reviewer for the study continuation.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Eugenia Ayrian, Associate Professor of Clinical Anesthesiology;Chief of Neuro Anesthesiology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-15-00615
Record Dates: First submitted 2017-03-29; First posted 2017-04-07 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Fusion of Spine, Lumbar Region
Keywords: Acetaminophen po; Acetaminophen IV; Pain management; minimally invasive lumbar fusions; Ofirmev; Analgesics; Opioid; Pain; Postoperative; Spinal
MeSH Terms: conditions — Agnosia; Pain | interventions — Acetaminophen; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetaminophen IV Soln 10 MG/ML (A) (Experimental): Patients in group A will receive 1 g of IV acetaminophen 15 minutes prior to wound incision, and every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Interventions: Drug: Acetaminophen IV Soln 10 MG/ML; Drug: Hydromorphone
- PO acetaminophen (B) (Experimental): Patients in group B will receive 1 g of PO acetaminophen prior to surgery, and 1 g of oral acetaminophen every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Interventions: Drug: Acetaminophen; Drug: Hydromorphone
- Hydromorphone (control arm) (C) (Active Comparator): Patients in the control arm (Group C) will not receive acetaminophen for 24 hours.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Acetaminophen IV Soln 10 MG/ML
  Other Names: Ofirmev
  Arms: Acetaminophen IV Soln 10 MG/ML (A)
Drug: Acetaminophen
  Other Names: Tylenol
  Arms: PO acetaminophen (B)
Drug: Hydromorphone
  Other Names: Dilaudid

SUMMARY:
Simple explanation and rationale:

Recovery after spine surgery is usually accompanied by severe pain which has traditionally been managed with opioids. It is common practice to supplement opioid treatment with different classes of analgesics which work through alternative pain pathways and receptors in order to achieve an additive or synergistic effect while reducing the amount of opioids necessary for pain control.

Acetaminophen can be a beneficial supplemental analgesic to opioids for postoperative pain relief.

Intervention:

Patients will be randomized to either the treatment with IV acetaminophen (A), PO acetaminophen (B), or hydromorphone control group (C).

Objective/Purpose:

Primary objective is to determine the impact of administering a supplemental non-opioid analgesic drug such as IV or PO acetaminophen on total opioid dose administered over the postoperative period.

Secondary objectives include investigating the impact of IV/PO acetaminophen on the level of postoperative pain, patient satisfaction, and side effects secondary to opioids such as nausea, vomiting, pruritus, sedation, respiratory depression, ileus, and urinary retention, and PACU (postoperative care unit) discharge time.

Study population:

126 patients will be enrolled in the study (42 for group A, 42 for group B, and 42 for control group C).

Follow-up and Endpoints / Outcomes:

Postoperative assessments will be done at 0, 30, and 60 minutes, 6 hours, 12 hours and 24 hours after surgery. Patients will be evaluated for pain (using a numeric rating scale), total opioid consumption, and for opioid side effects including drowsiness (using the Ramsey sedation scale and the Aldrete score at the time of arrival to and discharge from recovery room), respiratory depression, nausea, vomiting, and pruritus. Patient satisfaction will also be assessed using a numeric rating scale.

DETAILED DESCRIPTION:
Simple explanation and rationale:

Recovery after spine surgery, especially spinal fusion surgery, is usually accompanied by severe pain which has traditionally been managed with opioids. While opioids have been proven effective, they are associated with undesirable side effects including nausea, vomiting, pruritus, sedation, respiratory depression, ileus, and urinary retention leading to increased time required in recovery and a decrease in patient satisfaction. For this reason, it is common practice to supplement opioid treatment with different classes of analgesics which work through alternative pain pathways and receptors in order to achieve an additive or synergistic effect while reducing the amount of opioids necessary for pain control.

Acetaminophen is a centrally-acting cyclooxygenase inhibitor nonsteroidal anti-inflammatory medication that has minimal, if any, gastrointestinal and platelet-inhibiting side effects, and is better tolerated by patients than other cyclooxygenase inhibitors. This medication can be a beneficial supplemental analgesic to opioids for postoperative pain relief. Previously conducted studies demonstrate a rationale for the use of intravenous/PO acetaminophen in a multimodal analgesic regimen to reduce postoperative analgesia.

Intervention:

Patients will be randomized to either the treatment with IV acetaminophen (A), PO acetaminophen (B), or hydromorphone control group (C). Patients who are randomized to group A will receive 1 g of IV acetaminophen during the wound closure and every 4 to 6 hours postoperatively for a total of 4 g in 24 hours. Patients who are randomized to group B will receive 1 g of PO acetaminophen before surgery and every 4 to 6 hours postoperatively for a total of 4 g in 24 hours. Patients who are randomized to control group C will not receive acetaminophen. Post-operatively, patients in both groups will also receive IV hydromorphone PCA (patient-controlled analgesia) only for 24 hours for pain.

Objective/Purpose:

Primary objective is to determine the impact of administering a supplemental non-opioid analgesic drug such as IV or PO acetaminophen on total opioid dose administered over the postoperative period.

Secondary objectives include investigating the impact of IV/PO acetaminophen on the level of postoperative pain, patient satisfaction, and side effects secondary to opioids such as nausea, vomiting, pruritus, sedation, respiratory depression, ileus, and urinary retention, and PACU discharge time.

Study population:

126 patients will be enrolled in the study (42 for group A, 42 for group B, and 42 for control group C).

Follow-up and Endpoints / Outcomes:

Postoperative assessments will be done at 0, 30, and 60 minutes, 6 hours, 12 hours and 24 hours after surgery. Patients will be evaluated for pain (using a numeric rating scale), total opioid consumption, and for opioid side effects including drowsiness (using the Ramsey sedation scale and the Aldrete score at the time of arrival to and discharge from recovery room), respiratory depression, nausea, vomiting, and pruritus. Patient satisfaction will also be assessed using a numeric rating scale.

Statistics:

All sample size calculations with reference to:

* Specific Aim 1 reduction of opioid intake by at least 25% between the Control (Group C) and Intervention Groups A and B, and
* Specific Aim 2 improvement of Pain Score by at least 25% between the Control (Group C) and the Intervention Groups A and B,

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I-III patients scheduled for elective one or two level minimally invasive lumbar fusions

Exclusion Criteria:

* Patients requiring surgery for neoplastic processes
* Allergy to acetaminophen
* Liver dysfunction and elevated Liver Function Tests (LFTs)
* Alcohol or drug dependency
* Mental retardation
* Less than 50 kg of weight
* regnant women
* Patients requiring long-acting opioid pain management (including fentanyl patch, oxycontin, etc) for over 3 weeks immediately prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Ayrian, Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The data will kept for a minimum of 3 years after the study is completed. All documents containing identifiers will be shredded. Electronic documents will be deleted.

REFERENCES:
- [Background] Cakan T, Inan N, Culhaoglu S, Bakkal K, Basar H. Intravenous paracetamol improves the quality of postoperative analgesia but does not decrease narcotic requirements. J Neurosurg Anesthesiol. 2008 Jul;20(3):169-73. doi: 10.1097/ANA.0b013e3181705cfb. PMID 18580346
- [Background] Devin CJ, McGirt MJ. Best evidence in multimodal pain management in spine surgery and means of assessing postoperative pain and functional outcomes. J Clin Neurosci. 2015 Jun;22(6):930-8. doi: 10.1016/j.jocn.2015.01.003. Epub 2015 Mar 9. PMID 25766366
- [Background] Korkmaz Dilmen O, Tunali Y, Cakmakkaya OS, Yentur E, Tutuncu AC, Tureci E, Bahar M. Efficacy of intravenous paracetamol, metamizol and lornoxicam on postoperative pain and morphine consumption after lumbar disc surgery. Eur J Anaesthesiol. 2010 May;27(5):428-32. doi: 10.1097/EJA.0b013e32833731a4. PMID 20173643
- [Background] Garcia RM, Cassinelli EH, Messerschmitt PJ, Furey CG, Bohlman HH. A multimodal approach for postoperative pain management after lumbar decompression surgery: a prospective, randomized study. J Spinal Disord Tech. 2013 Aug;26(6):291-7. doi: 10.1097/BSD.0b013e318246b0a6. PMID 23887076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 patients were involved in study. 22 patients completed the study. Patients were recruited in the surgical clinic, preoperative clinic, preoperative surgical area.
Pre-assignment Details: Patients were included in the study according to their inclusion and exclusion criteria. There were no patients were excluded from study in the period after signing the consent to assignment to groups.
Groups:
- Acetaminophen IV Soln 10 Milligram/Milliliter (MG/ML) (A): Patients in group A will receive 1 g of IV acetaminophen 15 minutes prior to wound incision, and every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Acetaminophen IV Soln MG/ML
  Hydromorphone
- PO Acetaminophen (B): Patients in group B will receive 1 g of PO acetaminophen prior to surgery, and 1 g of oral acetaminophen every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Acetaminophen
  Hydromorphone
- Hydromorphone (Control Arm) (C): Patients in the control arm (Group C) will not receive acetaminophen for 24 hours.
  Hydromorphone
Period: Overall Study
Arm/Group | Acetaminophen IV Soln 10 Milligram/Milliliter (MG/ML) (A) | PO Acetaminophen (B) | Hydromorphone (Control Arm) (C)
Started | 11 | 11 | 6
Completed | 9 | 9 | 4
Not Completed | 2 | 2 | 2
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Acetaminophen IV Soln 10 MG/ML (A): Patients in group A will receive 1 g of IV acetaminophen 15 minutes prior to wound incision, and every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Acetaminophen IV Soln 10 MG/ML
  Hydromorphone
- Total: Total of all reporting groups
Arm/Group | Acetaminophen IV Soln 10 MG/ML (A) | PO Acetaminophen (B) | Hydromorphone (Control Arm) (C) | Total
Number analyzed (Participants) | 9 | 9 | 4 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 3 | 11
  >=65 years | 6 | 4 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 1 | 15
  Male | 4 | 0 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 8 | 7 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 4 | 22
Number of analyzed participants in each group [Count of Participants; unit: Participants] | 9 | 9 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Use
Description: Determine the impact of administering a supplemental non-opioid analgesic drug such as IV/oral acetaminophen on total opioid dose administered over the perioperative period.
Time Frame: Within 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Acetaminophen IV Soln 10 MG/ML (A): Hydromorphone and IV Acetaminophen are given to this group
- PO Acetaminophen (B): Hydromorphone and PO acetaminophen are given to this group
- Hydromorphone (Control Arm) (C): Hydromorphone only is given to the patients in this group
Arm/Group | Acetaminophen IV Soln 10 MG/ML (A) | PO Acetaminophen (B) | Hydromorphone (Control Arm) (C)
Number analyzed (Participants) | 9 | 9 | 4
mg
  PACU dose | 1.2 (0.4) | 1.3 (0.3) | 1.7 (0.5)
  Ward dose | 9.8 (2.9) | 10.4 (3.1) | 13 (5.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected within 24 hours.
Groups:
- Acetaminophen IV Soln 10 MG/ML (A): Patients in group A will receive 1 g of IV acetaminophen 15 minutes prior to wound incision, and every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Acetaminophen IV Soln 10 MG/ML
  Hydromorphone
  No adverse events.
- PO Acetaminophen (B): Patients in group B will receive 1 g of PO acetaminophen prior to surgery, and 1 g of oral acetaminophen every 4 to 6 hours postoperatively for a total of 4 grams in 24 hours.
  Acetaminophen
  Hydromorphone
  No adverse events.
- Hydromorphone (Control Arm) (C): Patients in the control arm (Group C) will not receive acetaminophen for 24 hours.
  Hydromorphone
  No adverse events.
Arm/Group | Acetaminophen IV Soln 10 MG/ML (A) | PO Acetaminophen (B) | Hydromorphone (Control Arm) (C)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/4

LIMITATIONS AND CAVEATS:
The trial was not completed and had very small amount of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03104816/Prot_SAP_000.pdf